CLINICAL TRIAL: NCT05975996
Title: Cyclophosphamide Added to Standard Immunosuppressive Therapy With Herombopag as Front-line Therapy in Patients With Severe Aplastic Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Fang Liwei, Associate Chief Physician of Regenerative Medical Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023038
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Severe Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiemental (Experimental): ALG/CsA(Cyclosporine) and herombopag and moderate-dose cyclophosphamide
  Interventions: Drug: Cyclophosphamide added to standard immunosuppressive therapy with herombopag

INTERVENTIONS:
Drug: Cyclophosphamide added to standard immunosuppressive therapy with herombopag — Severe aplastic anemia patients will receive a daily dose of Anti-lymphocyte globulin (25mg/kg) for the initial five days at the beginning of the treatment. Cyclosporine will be administered daily at a dosage of 3-5mg/kg. Herombopag will be administered daily at a dosage of 15mg starting from the first day of treatment and continuing for a duration of six months. The moderate-dose cyclophosphamide (20mg/kg) will be administered on days 29-30 and days 43-44.

SUMMARY:
This is a prospective, single-center, single-arm, phase 2 study. This study aims to evaluate the efficacy and safety of Anti-lymphocyte globulin plus herombopag in combination with moderate-dose cyclophosphamide for severe aplastic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 12 years
* Subject has a diagnosis of naïve severe or very severe aplastic anemia
* ECOG performance status ≤2
* Unwilling or unable to receive allogeneic hematopoietic stem cell transplantation.
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Previously received immunosuppressive therapy > 4 weeks
* Previously treated with TPO-RA > 4 weeks
* Have an allergy or intolerance to either herombopag or cyclophosphamide.
* Have an allergy to ALG
* Uncontrolled systemic fungal, bacterial, or viral infection
* Poorly controlled hypertension (≥140/90mmHg) or diabetes (a fasting plasma glucose concentration ≥7.0mmol/L or a random venous plasma glucose concentration ≥11.1mmol/L)
* Abnormal liver or kidney function: ALT or AST >3 ULN, or serum creatinine (sCr)≥ 2.5 ULN.
* History of radiotherapy and chemotherapy for malignant solid tumors
* Combined with other serious disorders
* Pregnant or breast-feeding patients
* Patients considered to be ineligible for the study by the investigator for reasons other than the above.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Within 3 months
  Percentage of patients with hematological response. Hematological response includes complete rate, near complete rate(CR), very good partial response(VGPR), good partial response(GPR) and partial response(PR).

SECONDARY OUTCOMES:
Robust response | Within 3 months
  Percentage of patients with robust response, including CR, near CR, VGPR and GPR.
All-cause mortality | Within 3 months
Time to achieve robust hematological response | Within 6 months
Incidence of the adverse event | Within 6 months
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Fang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China